CLINICAL TRIAL: NCT00000400
Title: Bone Formation-Resorption Coupling and Osteoporosis
Brief Title: Alendronate and/or Parathyroid Hormone for Osteoporosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Robert M. Neer, MD, Physician, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P50 AR44855 NIAMS-023; P50AR044855 (NIH)
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2013-12

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; Bone formation; Bone resorption; Parathyroid hormone (PTH); Postmenopause
MeSH Terms: conditions — Osteoporosis; Bone Resorption | interventions — PTH protein, human; Teriparatide; Alendronate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PTH (Experimental): Human parathyroid hormone [hPTH-(1-34)]
  Interventions: Drug: Human parathyroid hormone [hPTH-(1-34)]
- ALN (Active Comparator): Alendronate
  Interventions: Drug: alendronate
- PTH+ALN (Experimental): Human parathyroid hormone [hPTH-(1-34)] plus alendronate
  Interventions: Drug: Human parathyroid hormone [hPTH-(1-34)]; Drug: alendronate

INTERVENTIONS:
Drug: Human parathyroid hormone [hPTH-(1-34)] — 37 mcg once daily by self-administered sc injection
  Other Names: teriparatide
  Arms: PTH; PTH+ALN
Drug: alendronate — 70 mg/week by oral route
  Other Names: Fosamax
  Arms: ALN; PTH+ALN

SUMMARY:
This study looks at the effects of two medications, alendronate and parathyroid hormone, on bone mass and on bone formation and bone breakdown in women with osteoporosis. We will randomly select postmenopausal women who have osteoporosis to receive laboratory-produced human parathyroid hormone (hPTH), or alendronate, or both for 2.5 years. Study participants will return to the study center periodically to have their bone mass measured and to give blood and urine samples for tests of bone formation and breakdown and for other laboratory tests. Those who complete the study are eligible for one or two 12 month extension studies.

DETAILED DESCRIPTION:
This is a randomized, prospective, open-label study in which osteoporotic postmenopausal women self-administer synthetic hPTH-(1-34), alendronate, or both, every day for 2.5 years. Participants initially come to Massachusetts General Hospital once a month, and subsequently once every 3-6 months, for measurements of serum and urine indices of bone formation and resorption, serum and urine toxicity tests, and DXA/QCT measurements of bone mass. One-third of the participants take hPTH-(1-34) daily, one-third take alendronate once daily, and one-third take both daily (Phase A, months 0-30).

Participants who complete Phase A are eligible for a 12 month extension study (Phase B, months 30-42), during which any alendronate treatment is continued without change and any hPTH 1-34 treatment is stopped.

Participants who complete Phase B are eligible for a second 12 month extension study (Phase C, months 42-54), during which any alendronate treatment is continued without change and every participant takes hPTH 1-34.

During Phases B and C, these participants come to Massachusetts General Hospital once every 6 months for measurements of serum and urine indices of bone formation and resorption, serum and urine toxicity tests, and DXA/QCT measurements of bone mass.

ELIGIBILITY:
Inclusion Criteria:

* Lumbar spine or hip BMD T-score less than or equal to minus 2.0
* Postmenopausal at least 5 years
* Fully ambulatory
* Able to give informed consent

Exclusion Criteria:

* No concurrent illnesses that cause bone loss
* No recent drug treatment for osteoporosis
* No recent fracture

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 1999-08; Primary Completion 2006-04 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
change in spine bone mineral density | study months 30 (phase A), 42 (phase B), 54 (phase C)

SECONDARY OUTCOMES:
change in hip bone mineral density | study months 30 (phase A), 42 (phase B), 54 (phase C)
change in forearm bone mineral density | study months 30 (phase A), 42 (phase B), 54 (phase C)
change in total body bone mineral | study months 30 (phase A), 42 (phase B), 54 (phase C)
change in femoral shaft bone mineral density | study months 30 (phase A), 42 (phase B), 54 (phase C)
change in serum PINP | study months 0-30 (phase A), 30-42 (phase B), 42-54 (phase C)
change in serum osteocalcin | study months 0-30 (phase A), 30-42 (phase B), 42-54 (phase C)
change in serum NTX | study months 0-30 (phase A), 30-42 (phase B), 42-54 (phase C)
incidence of hypercalcemia | study months 0-30 (phase A), 30-42 (phase B), 42-54 (phase C)
incidence of hypercalciuria | study months 0-30 (phase A), 30-42 (phase B), 42-54 (phase C)
incidence of symptoms | study months 0-30 (phase A), 30-42 (phase B), 42-54 (phase C)

CONTACTS AND LOCATIONS:
Overall Officials: Robert M. Neer, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Finkelstein JS, Wyland JJ, Leder BZ, Burnett-Bowie SM, Lee H, Juppner H, Neer RM. Effects of teriparatide retreatment in osteoporotic men and women. J Clin Endocrinol Metab. 2009 Jul;94(7):2495-501. doi: 10.1210/jc.2009-0154. Epub 2009 Apr 28. PMID 19401368
- See also: Click here for more information about this study. — http://www.mgh.harvard.edu